CLINICAL TRIAL: NCT04189939
Title: Computational Psychiatric Approach for Prognosis of Medication-Resistant Depression
Brief Title: Computational Psychiatric Approach to Depression
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00056131
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-10

CONDITIONS: Depression; Treatment Resistant Depression
Keywords: ECT treatment; treatment-resistant depression; neural changes
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- subjects with treatment-resistant depression: approximately 48 subjects with treatment-resistant depression will undergo (1) clinical assessments, (2) perform a computer-based decision-making task while (3) their brain activity is monitored using a 3T MRI scanner.
  Interventions: Other: clinical assessments
- healthy subjects: approximately 48 healthy subjects will undergo (1) clinical assessments, (2) perform a computer-based decision-making task while (3) their brain activity is monitored using a 3T MRI scanner.
- subjects with non treatment-resistant depression: approximately 48 subjects with non-treatment-resistant depression will undergo (1) clinical assessments, (2) perform a computer-based decision-making task while (3) their brain activity is monitored using a 3T MRI scanner.

INTERVENTIONS:
Other: clinical assessments — Behavioral tasks will be executed via a computer interface. Below, we provide an estimated timeline for each visit and subsequently provide detail for the relevant stages.
  Each participant's visit will last approximately 4-5 hours. Each visit will consist of the following tasks (in this order):
  Other Names: computer-based decition making task; 3T MRI scan
  Groups: subjects with treatment-resistant depression

SUMMARY:
The purpose of this research is to investigate how the brain changes in patients undergoing electroconvulsive (ECT) treatment for depression. Subjects will be invited to be in this study because (1) they are a patient about to receive ECT treatment for depression, or (2) they are a patient diagnosed with depression and do not qualify for ECT treatment, or (3) they are a healthy adult volunteer with no history of depression.

All volunteers must be between the ages of 18-85. Participation in this research will involve three visits. Each visit will last about 3-4 hours. If the subject is a patient receiving ECT for depression the study team will schedule study visits to go along with patient treatment visits. If the subject is diagnosed with depression (not treatment-resistant depression) or are a healthy volunteer, their first visit will be scheduled at their convenience, followed by a second visit 1-3 months post visit one and a third visit 1-2 months post visit two, for a total of three research visits.

Participation in this research will involve playing simple computer games while the subject's brain is scanned with magnetic resonance imaging (MRI). Additionally, the study team will assess symptoms of depression using questionnaires. Patients receiving ECT will not experience any changes to their standard of care ECT treatment plan. Healthy and non-treatment resistant depressed volunteers will not undergo ECT treatment.

DETAILED DESCRIPTION:
The goal for this study will be to test the following overall hypotheses: (1) that adaptive decision-making processes are disrupted in patients with treatment-resistant depression, and (2) the neural and behavioral changes associated with treatment-resistant depression can be assessed using functional magnetic resonance imaging paired with computationally constrained adaptive decision-making games.

The investigators will use computational modeling of incentivized decision-making tasks, brain imaging (functional magnetic resonance imaging, fMRI), and standard clinical assessments, to characterize patients referred to Wake Forest Baptist Medical Center for ECT. Characterization will occur over multiple visits to be aligned with the normal course of patient care.

Data collected may be used in hypothesis driven analyses to:

1. classify treatment resistant depression versus healthy controls and non-treatment resistant depression
2. predictors of ECT treatment success versus failure
3. characterize brain and behavioral changes consistent with treatment success versus failure
4. predict who will need maintenance ECT therapy
5. determine what changes in decision-making behavior are apparent in patients who require ECT maintenance therapy versus those who do not.

ELIGIBILITY:
For patients:

Inclusion Criteria:

* Adult volunteers (ages 18-85)
* Treatment-resistant depressed patients must meet criteria in standard-of-care evaluation for ECT treatment
* Clinically depressed patients must meet criteria in standard-of-care evaluation for depression.

Exclusion Criteria:

* Individuals who cannot have MRI scanning
* Individuals not able to provide written consent and verbal assent
* Individuals not able to understand task instructions or consent documents
* Women who are pregnant

For healthy subject volunteers:

Inclusion Criteria:

* Healthy adult volunteers (ages 18-85)

Exclusion Criteria:

* Individuals diagnosed with depression (regardless of treatment status)
* Individuals who cannot have MRI scanning
* Individuals not able to provide written consent and verbal assent
* Individuals not able to understand task instructions or consent documents
* Women who are pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet the criteria in standard-of-care evaluation for ECT treatment, clinically depressed patients (non-treatment-resistant), and healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Functional Brain scanning - Neural activation | Baseline
  neural activation measured during functional MRI
Functional Brain scanning - Neural activation | month 1
  neural activation measured during functional MRI
Functional Brain scanning - Neural activation | month 2
  neural activation measured during functional MRI

SECONDARY OUTCOMES:
Sensation Seeking Scale | Baseline, month 1, month 2
  This scale is a 43-item. Total score 0-430, higher number denotes worse outcomes.
Perceived Control of Internal States Scale (PCISS) | Baseline, month 1, month 2
  The PCISS is an 18-item scale designed to measure respondents' perceptions of their ability to control their internal states and to moderate the impact of aversive events on their emotions, thoughts and physical well-being. Scores can range from 18 to 90, with high scores indicating higher levels of perceived control of internal states.
Montreal Cognitive Assessment | Baseline, month 1, month 2
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment.MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal, the lower number denotes worse outcomes.
Physical Risk Assessment Inventory | Baseline, month 1, month 2
  27 Items. Total score 0- 162, higher number denotes worse outcomes.
Patient Health Questionnaire-9 | Baseline, month 1, month 2
  The Patient Health Questionnaire (PHQ) is an instrument for making criteria-based diagnoses of depressive disorders commonly. Total score 1-29, higher scores denote worse severity of depression.
Hamilton Depression Inventory (HAM-D) | Baseline, month 1, month 2
  The HAM-D is designed to rate the severity of depression in patients. Total score 0-54, higher scores denote worse severity of depression.

OTHER OUTCOMES:
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, month 1, month 2
  The SHAPS is a self-administered questionnaire with 14 items assessing domains of pleasure response/hedonic experience. Total score ranges from 0-42 with higher scores indicating increased anhedonia.
Positive Valence Systems Scale (PVSS) | Baseline, month 1, month 2
  The PVSS is a self-administered 21-item questionnaire measuring the NIMH's Research Domain Criteria Positive Valence System Domain. Total score ranges from 1-189, with higher scores denoting increased response to rewards.
Columbia Suicide Scale (C-SSRS) | Baseline, month 1, month 2
  The C-SSRS is designed to rate an individual's risk for suicide based on lifetime and recent ideations. Scores can range from no risk, low risk, moderate risk, and high risk.
Apathy Motivation Index (AMI) | Baseline, month 1, month 2
  The AMI is an 18-item self-report index of apathy and motivation in Behavioral, Social, and Emotional Domains. Total score in each domain is 0-24 with higher scores denoting increased apathy.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth T Kishida, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kishida KT, King-Casas B, Montague PR. Neuroeconomic approaches to mental disorders. Neuron. 2010 Aug 26;67(4):543-54. doi: 10.1016/j.neuron.2010.07.021. PMID 20797532
- [Background] Montague PR, Dolan RJ, Friston KJ, Dayan P. Computational psychiatry. Trends Cogn Sci. 2012 Jan;16(1):72-80. doi: 10.1016/j.tics.2011.11.018. Epub 2011 Dec 14. PMID 22177032
- [Background] Wang XJ, Krystal JH. Computational psychiatry. Neuron. 2014 Nov 5;84(3):638-54. doi: 10.1016/j.neuron.2014.10.018. Epub 2014 Nov 5. PMID 25442941
- [Background] Huys QJ, Maia TV, Frank MJ. Computational psychiatry as a bridge from neuroscience to clinical applications. Nat Neurosci. 2016 Mar;19(3):404-13. doi: 10.1038/nn.4238. PMID 26906507
- [Background] Berlim MT, Turecki G. Definition, assessment, and staging of treatment-resistant refractory major depression: a review of current concepts and methods. Can J Psychiatry. 2007 Jan;52(1):46-54. doi: 10.1177/070674370705200108. PMID 17444078